CLINICAL TRIAL: NCT05839743
Title: Investigation of the Effects of Aerobic Exercise, Balance Exercise and Combined Exercise Practices on Frailty, Balance, Fall Risk, Reaction Time, Cognitive Functions and Quality of Life in Dementia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Ilkem Guzel, Lecturer, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24032023
Record Dates: First submitted 2023-04-03; First posted 2023-05-03 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Dementia; Aerobic Exercise; Balance Exercise; Cognitive Function; Frailty; Reaction Time
MeSH Terms: conditions — Dementia; Frailty | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Group (Experimental)
  Interventions: Other: Aerobic Exercise
- Balance Exercise Group (Experimental)
  Interventions: Other: Balance Exercise
- Combined Exercise Group (Experimental)
  Interventions: Other: Combined Exercise

INTERVENTIONS:
Other: Aerobic Exercise — The aerobic exercise program will be specially prepared for the participants and will aim to rhythmically exercise large muscle groups. The exercise will be performed twice a week for 6 weeks at 50-75% of maximum heart rate for 20-50 minutes per session. Each exercise will last 30-60 minutes in total, after adding 5 minutes of warm-up and 5 minutes of cool-down before and after the exercise. The participant's pulse will be monitored continuously during the exercise.
  Arms: Aerobic Exercise Group
Other: Balance Exercise — Balance exercises belonging to the Otago Exercise Program and other balance exercises used in the elderly will be prepared specifically for the participant and will be applied 2 days a week for 6 weeks in combination. Before and after the exercise, a 5-minute warm-up and 5-minute cool-down exercise will be performed.
  Arms: Balance Exercise Group
Other: Combined Exercise — In the combined exercise program, first balance exercises and then aerobic exercise program will be applied 2 days a week for 6 weeks.
  Arms: Combined Exercise Group

SUMMARY:
Dementia is a clinical disorder characterized by progressive and permanent loss of multiple cognitive functions, especially memory, at a level that affects activities of daily living. There is no pharmacologic treatment method that can change the prognosis in dementia. The methods used today are symptomatic and cause various side effects. For this reason, non-pharmacologic approaches are on the agenda in the treatment of dementia. Among these approaches, physical activity approaches such as symptomatic treatment or exercise come to the forefront due to their prognosis-slowing effects. There are also many studies showing that dementia is directly related to physical performance and frailty. Deterioration of physical performance, increased frailty, and decreased muscle strength create a vicious circle with the prognosis of dementia. In addition, patients with dementia have balance problems due to prolonged reaction time, cognitive impairment and physical problems, and the risk of falls increases. In order to prevent the risk of falls, exercise practices are of great importance. Although the effects of aerobic exercise on dementia have been examined many times in the literature, there are very few studies examining the effects of balance exercises and combined exercises. In addition, physical characteristics such as frailty and muscle weakness, which are very common in patients with dementia, have not been evaluated as a whole in studies on patients with dementia. Therefore, this study will be conducted to comparatively examine the effects of combined aerobic exercise and balance exercises on balance and falls, frailty, muscle strength, cognitive functions, and reaction time in patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years,
* To be able to speak and understand Turkish,
* To have at least primary education,
* Perceive and adapt to simple commands,
* Scoring between 18-23 on the standardized mini mental state assessment scale (200),
* To be able to provide independent mobilization,
* Volunteering to participate.

Exclusion Criteria:

* Rapid progression of dementia (infectious, vascular, hematologic diseases),
* Cardiac or cerebrovascular event, endocrine disorder, fluid-electrolyte imbalance or infection during the follow-up period,
* Presence of malignancy,
* Detection of a delirium picture,
* Presence of severe depression,
* Participate in a regular exercise program for at least 6 months before the study,
* Having a fracture or fracture surgery in the lower extremity within the last year,
* Any orthopedic problem that prevents him/her from exercising.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Edmonton Frailty Scale | Change from Baseline Edmonton Frailty Scale at 6 weeks
  0 - 5 = Not Frail, 6 - 7 = Vulnerable, 8 - 9 = Mild Frailty, 10-11 = Moderate Frailty, 12-17 = Severe Frailty
Muscle Strength Assessment for Sarcopenia | Change from Baseline Muscle Strength Assessment for Sarcopenia at 6 weeks
  Muscle strength measurement in kg with a dynamometer
30 Seconds Sit To Stand Test | Change from Baseline 30 Seconds Sit To Stand Test at 6 weeks
  For testing leg strength and endurance in older adults. The score is the total number of stands within 30 seconds.
Single Leg Stance Test | Change from Baseline Single Leg Stance Test at 6 weeks
  If unable to stand for 5 seconds or less client at greater risk of injury from fall.
Tinetti Balance and Gait Assessment | Change from Baseline Tinetti Balance and Gait Assessment at 6 weeks
  The Tinetti test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling.
Dynamic Gait Index | Change from Baseline Dynamic Gait Index at 6 weeks
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score on the Dynamic Gait Index is a 24.
Functional Reach Test | Change from Baseline Functional Reach Test at 6 weeks
  10"/25 cm or greater Low risk of falls; 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal; 6"/15cm or less Risk of falling is 4x greater than normal; Unwilling to reach Risk of falling is 8x greater than normal.
Johns Hopkins Fall Risk Assessment Tool | Change from Baseline Johns Hopkins Fall Risk Assessment Tool at 6 weeks
  6-13 Total Points = Moderate Fall Risk, >13 Total Points = High Fall Risk
Reaction Time Test | Change from Baseline at 6 weeks
  The 3 reaction times recorded in milliseconds are averaged.
Mini Mental State Examination | Change from Baseline Reaction Time Test at 6 weeks
  The maximum score for the Mini Mental State Examination is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
The World Health Organization Quality of Life - Old Module | Change from Baseline The World Health Organization Quality of Life - Old Module at 6 weeks
  It is scored in the range of 4-20. The higher the score, the better the quality of life.
Geriatric Depression Scale | Change from Baseline Geriatric Depression Scale at 6 weeks
  There are 15 questions. Each question is worth 1 point. A score of 5 or more suggests depression.
Wechsler Memory Scale | Change from Baseline Wechsler Memory Scale at 6 weeks
  Scored on 1-19 Scaled Score Metric. High scores (13 and above) indicate better than expected performance on the dependent variable given performance on the control variable. Low scores (7 and below) indicate poorer than expected performance on the dependent score given performance on the control score. Scores in the average range (8-12) indicate no difference in performance between the control and dependent measures.
Mental Rotation Test | Change from Baseline Mental Rotation Test at 6 weeks
  Contains 20 pairs of items worth 1 point each. A high score indicates good mental rotation skill.
Spatial Orientation Test | Change from Baseline Spatial Orientation Test at 6 weeks
  Contains 20 pairs of items worth 1 point each. A high score indicates good spatial orientation skill.

CONTACTS AND LOCATIONS:
Locations (1):
- Ihlamur Konağı Nursing Home and Elderly Care Center, Ankara, Çankaya, Turkey (Türkiye)